CLINICAL TRIAL: NCT00837434
Title: A Partially Blinded, Randomized, Multi-Center, Phase IV Trial to Evaluate Mechanism of Action of Anti-TNF Agents in Rheumatoid Arthritis
Brief Title: Anti-TNF Agents for the Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAIT ARA06; NIAID CRMS ID#: 20001 (Other: DAIT NIAID)
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Results first posted 2015-04-14 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Rheumatoid Arthritis
Keywords: tumor necrosis factor (TNF) blockade; inflammatory autoimmune disorder
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Adalimumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etanercept (Experimental): Participants receive a subcutaneous injection of etanercept once every week for 24 weeks
  Interventions: Drug: Etanercept
- Adalimumab (Experimental): Participants receive a subcutaneous injection of adalimumab once every 2 weeks for 24 weeks
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Etanercept — 50 mg dose of etanercept by subcutaneous injection
  Other Names: Enbrel®
  Arms: Etanercept
Drug: Adalimumab — 40 mg dose of adalimumab by subcutaneous injection
  Other Names: Humira®)
  Arms: Adalimumab

SUMMARY:
Rheumatoid arthritis (RA) is a chronic disease that leads to inflammation and progressive joint damage. RA is a systemic inflammatory autoimmune disorder affecting almost 1% of the United States population. Current therapies target the immune system early in the disease process before joint damage occurs, and include drugs such as methotrexate (MTX) and tumor necrosis factor (TNF)-blocking agents. The primary purpose of this study is to determine the effectiveness of two TNF inhibitors, etanercept and adalimumab, on memory B lymphocytes (B-cells) in the peripheral blood of participants with RA.

Additionally, there are 4 optional sub-studies as part of the trial:

* B-Cell Kinetic Sub-Study to look at changes in B-cell subsets over time and how quickly reductions in B-cell memory occur
* Vaccine Response Sub-Study to assess B cell memory in response to immunization with hepatitis B,-hepatitis A, and diphtheria/tetanus vaccines, and to determine whether T-cell vaccine responses are altered with TNF blockade
* Tonsil Biopsy Sub-Study to evaluate how TNF blockade affects memory B-cells in the tonsil dendritic cells and germinal cells
* Synovial Biopsy Sub-Study to evaluate how TNF blockade affects changes in memory B-cells in lymphoid tissue.

DETAILED DESCRIPTION:
RA is characterized by persistent inflammation of peripheral joints, causing pain, stiffness, swelling and warmth. Over the past 10 years, advancements in biotechnology have revolutionized RA therapeutics with biologically-derived immunomodulating compounds. TNF-alpha inhibitors constitute the largest class of these new biologic therapies. The purpose of this study is to determine the effectiveness two TNF inhibitors, etanercept and adalimumab, on memory B lymphocytes (B-cells) in the peripheral blood of participants with RA.

This study will last 24 weeks. Participants will be randomized into one of two treatment groups. Participants in one group will receive a dose of etanercept once every week for 24 weeks. Participants in the other group will receive a dose of adalimumab once every 2 weeks for 24 weeks.

This study consists of seven study visits after randomization and will occur at study entry and Weeks 4, 8, 12, 16, 20 and 24. Blood collection will occur at all study visits. A written participant assessment, vital signs, and physical exam will occur at study entry and Weeks 12 and 24. Follow-up calls to assess safety are scheduled for Weeks 4, 8, 16, and 20.

Additionally, participants will be offered the opportunity to enter one of four sub-studies as mentioned in the brief summary above: B Cell Kinetic Sub-Study, Vaccine Response Sub-Study, Tonsil Biopsy Sub-Study, and Synovial Biopsy Sub-Study. More information on these sub-studies is in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA*
* Disease duration as defined from the onset of symptoms of at least 3 months prior to study entry
* Active RA with DAS28 > 4.4, clinically requiring the addition of anti-TNF therapy
* Stable dose of MTX between 7.5 mg and 25 mg weekly for at least 8 weeks prior to study entry
* Able and willing to self-administer subcutaneous injections or have available qualified person(s) or caregiver to administer subcutaneous injections
* For females, agree to use accepted methods of contraception during the duration of the study and for 150 days after study completion*. *More information on these criterion can be found in the protocol.

Exclusion Criteria:

* Positive PPD test - a tuberculosis (TB) skin test: (> 5 mm induration regardless of prior Bacille Calmette-Guerin [BCG] vaccine administration) without evidence of ongoing treatment for at least 30 days or completed treatment
* History of positive PPD or chest x-ray findings indicative of prior TB infection, without documentation of either treatment for TB infection or chemoprophylaxis for TB exposure
* Prednisone dose > 10 mg/day (or equivalent dose of another corticosteroid) within 30 days prior to study entry
* Definitive diagnosis of another autoimmune disease that may require immunosuppression for treatment*
* Concomitant use of DMARDSs (e.g., disease-modifying antirheumatic drugs)*
* Any immunosuppressive therapy other than MTX, NSAIDs, or corticosteroids*
* Current or previous use of any biologic agent
* Presence of open leg ulcers
* Chronic or persistent infection that might be worsened by immunosuppressive treatment*
* Active infection or severe infections requiring hospitalization or treatment with intravenous (IV) antibiotics, IV antivirals, or IV antifungals within 30 days prior to study entry
* Received oral antibiotics, antivirals, or antifungals within 14 days prior to study entry
* Certain abnormal laboratory values*
* Any medical condition that, in the opinion of the investigator, would interfere with the study
* History of malignancy other than treated localized carcinoma in situ of the cervix or adequately treated non-metastatic squamous or basal cell skin carcinoma within 10 years prior to study entry
* Any Investigational agent within the earlier of 4 weeks or 5 half-lives prior to study entry
* History of drug or alcohol abuse within 6 months prior to study entry
* Known allergy or hypersensitivity to study products
* Inability or unwillingness to follow the protocol
* Any condition or treatment that, in the opinion of the investigator, places the participant at an unacceptable risk
* Pregnant or breastfeeding *More information on these criterion are in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-03; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A. Anolik, MD, PhD, Study Chair — University of Rochester; Inaki Sanz, MD, Study Chair — University of Rochester; R. John Looney, MD, Study Chair — University of Rochester; Meggan Mackay, MD, Principal Investigator — The Feinstein Institute for Medical Research NS-LIJ Health System; Jeffrey Curtis, MD, Principal Investigator — University of Alabama at Birmingham
Locations (7):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Yale University School Medicine, New Haven, Connecticut
  - University of Chicago, Chicago, Illinois
  - Feinstein Institute for Medical Research, Manhasset, New York
  - University of Rochester, Rochester, New York
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- [Background] Bingham CO 3rd. Emerging therapeutics for rheumatoid arthritis. Bull NYU Hosp Jt Dis. 2008;66(3):210-5. PMID 18937634
- [Background] Otomo K, Koike T. [TNF inhibitors for treatment of rheumatoid arthritis]. Nihon Naika Gakkai Zasshi. 2008 Oct 10;97(10):2405-12. doi: 10.2169/naika.97.2405. No abstract available. Japanese. PMID 19149036
- [Background] Soen S. [Daily practice using the guidelines for prevention and treatment of osteoporosis. The effects of anti-TNF therapy on bone and joint manifestations in rheumatoid arthritis]. Clin Calcium. 2008 Aug;18(8):1169-75. Japanese. PMID 18677056
- [Result] Meednu N, Barnard J, Callahan K, Coca A, Marston B, Thiele R, Tabechian D, Bolster M, Curtis J, Mackay M, Graf J, Keating R, Smith E, Boyle K, Keyes-Elstein L, Welch B, Goldmuntz E, Anolik JH. Activated Peripheral Blood B Cells in Rheumatoid Arthritis and Their Relationship to Anti-Tumor Necrosis Factor Treatment and Response: A Randomized Clinical Trial of the Effects of Anti-Tumor Necrosis Factor on B Cells. Arthritis Rheumatol. 2022 Feb;74(2):200-211. doi: 10.1002/art.41941. Epub 2021 Dec 27. PMID 34347945
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY824 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY824 — The Immunology Database and Analysis Portal (ImmPort) is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts. The portal includes available analysis tools for researchers.
- Available data/document: Study Protocol: SDY824 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY824 — ImmPort study identifier is SDY824.
- Available data/document: Study summary, -design, -adverse event(s), -summary of participant assessments, -medications, -demographics, -lab tests, -mechanistic assays, -study files et al.: SDY824 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY824 — ImmPort study identifier is SDY824.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were to be recruited from seven sites in the United States. Recruitment occurred at six sites. The first site was activated in April 2009. The first participant was randomized in July 2009 and the last participant was randomized in July 2013.
Groups:
- Etanercept: Participants were randomized to receive 50 mg etanercept given by subcutaneous injection every week for 24 weeks.
- Adalimumab: Participants were randomized to receive one subcutaneous injection of 40 mg adalimumab every other week for 24 weeks.
Period: Overall Study
Arm/Group | Etanercept | Adalimumab
Started | 43 | 20
Completed | 34 | 19
Not Completed | 9 | 1
Not completed — Physician Decision | 3 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawn by sponsor/regulatory agency | 1 | 0
Not completed — Noncompliant | 2 | 0
Not completed — Baseline assessments not done in time | 1 | 0
Not completed — Unable to obtain study drug | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Modified Intent-to-Treat population included all randomized subjects who received at least one dose of either etanercept or adalimumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept | Adalimumab | Total
Number analyzed (Participants) | 39 | 19 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (9.4) | 52.7 (14.0) | 52.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 15 | 46
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 9
  Not Hispanic or Latino | 31 | 18 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 30 | 18 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 39 | 19 | 58
Detection of Either IgM-Rheumatoid Factor or Antibodies to Cyclic Citrullinated Peptide [Number; unit: participants] — Serum IgM-Rheumatoid Factor (IgM RF) is an antibody often present in the blood of a person with rheumatoid arthritis. Positive value for RF: >/=0.5 IU/mL. Negative value for RF: <0.5 IU/mL. Presence of IgM RF indicates aggressive rheumatoid arthritis (RA) and higher risk of joint damage. Antibodies to Cyclic Citrullinated Peptide (anti-CCP) is often detected in in the blood of individuals with RA. Positive value for anti-CCP: >/=8 IU/mL. Negative value for anti-CCP: <8 IU/mL. High anti-CCP indicates an aggressive RA and a higher risk of joint damage.
  participants
    Positive | 30 | 14 | 44
    Negative | 9 | 5 | 14
Detection of IgM-Rheumatoid Factor (IgM RF) [Number; unit: participants] — Serum IgM RF is an antibody often present in the blood of a person with rheumatoid arthritis. Positive value for RF: >/=0.5 IU/mL. Negative value for RF: <0.5 IU/mL. Presence of IgM RF indicates aggressive rheumatoid arthritis (RA) and higher risk of joint damage.
  participants
    Positive | 24 | 9 | 33
    Negative | 15 | 10 | 25
Detection of Antibodies to Cyclic Citrullinated Antibody Peptide [Number; unit: participants] — Anti-CCP is often present in the blood of individuals with RA. Positive value for anti-CCP: >/=8 IU/mL. Negative value for anti-CCP: <8 IU/mL. High anti-CCP indicates an aggressive RA and a higher risk of joint damage.
  participants
    Positive | 25 | 11 | 36
    Negative | 14 | 8 | 22
Methotrexate Dosage [Mean (Standard Deviation); unit: mg] — Participants were required to be on a stable dose of methotrexate to be enrolled in the study. Stable dose definition: between 7.5 mg and 25 mg by mouth or subcutaneously weekly for at least 8 weeks prior to randomization.
  mg | 17.4 (4.0) | 18.8 (3.8) | 17.9 (3.9)
Years with Rheumatoid Arthritis [Mean (Standard Deviation); unit: years] — Years since diagnosis of rheumatoid arthritis by a physician. Participants were required to be diagnosed with Rheumatoid Arthritis at least 3 months before enrolling in the study.
  years | 5.8 (7.7) | 4.3 (5.2) | 5.3 (7.0)
Health Assessment Questionnaire-Disability Index (HAQ-DI) Score [Mean (Standard Deviation); unit: scores on a scale] — HAQ-DI is derived based on the mean of individual scores in 8 categories of daily living activities (using 20 questions). Each question is scored 0-3 (0=no difficulty, 1=some difficulty, 2=much difficulty, and 3=unable to do). In addition, category scores are modified if an aid or device is used, for example, a walker, or help is received from another person in the daily living activities. Scores from each of the 8 categories are totaled and can range from 0 to 24.
  scores on a scale | 1.4 (0.7) | 1.3 (0.6) | 1.4 (0.7)
C-reactive Protein (CRP) Level [Mean (Standard Deviation); unit: mg/L] — CRP is an acute phase reactant that is used to identify the presence of nonspecific inflammation. The CRP normal reference range depends on the laboratory. In this study the upper limit of normal ranged from 4 to 10.9 mg/L. An increased CRP level indicated the presence of inflammation. A low CRP may mean an absence of inflammation.
  mg/L | 14.1 (25.5) | 13.3 (24.3) | 13.8 (24.9)
Tender Joint Count [Mean (Standard Deviation); unit: Joints] — Tender Joint Count (TJC) is calculated based on tenderness response of 28 joints examined. TJC possible values range from 0 to 28. A lower TJC indicates less joint tenderness.
  Joints | 12.2 (6.6) | 12.6 (7.2) | 12.3 (6.7)
Swollen Joint Count at Baseline [Mean (Standard Deviation); unit: Joints] — Swollen Joint Count (SJC) is calculated based on swelling response of 28 joints examined. SJC possible values range from 0 to 28. A lower SJC indicates less joint swelling.
  Joints | 9.9 (6.2) | 9.4 (5.9) | 9.7 (6.0)
Patient's Global Assessment of Disease Activity- Visual Analog Scale (PtGADA-VAS) [Mean (Standard Deviation); unit: cm] — A self-reported measure of perceived disease activity obtained by responding to the question "considering all the ways that your arthritis affects you, rate how you are doing on the following scale by placing a vertical mark." A vertical mark on a 10 cm line rated 0 (very well) to 10 (very bad) determines the score. The range: 0 to 10, with 10 being severe symptoms).
  cm | 5.9 (2.6) | 7.3 (2.0) | 6.4 (2.5)
Disease Activity Score Using C-reactive Protein (DAS28-CRP) [Mean (Standard Deviation); unit: scores on a scale] — The DAS28 is: a score on a scale (0 to 10) indicating current activity of rheumatoid arthritis (>5.1=high disease activity; <=3.2=low disease activity; <2.6=remission); a continuous variable which is a composite of 4 variables(the number of tender joints out of 28, the number of swollen joints out of 28 joints, serum C-reactive protein (CRP) in mg/L and subject assessment of disease activity measure on a visual analogue scale (VAS) of 100 mm).
  scores on a scale | 5.2 (1.0) | 5.4 (0.7) | 5.3 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of CD27+ Switched Memory B Cells at Week 12
Description: Analysis of the steady state composition of the B cell compartment were performed using ex-vivo multicolor flow cytometry on Ficoll isolated peripheral blood mononuclear cells (PBMCs). CD27+ switched memory B cells are a subset of B cells and are assessed by flow cytometry. CD27+ switched memory B cells are expressed as a percent of B cells. Lower CD27+ memory B cells indicate a decrease in the generation of B cell memory which may be caused by blocking lymphotoxin (LT) and tumor necrosis factor (TNF) signaling.
Time Frame: Week 12
Population: The Per Protocol population includes subjects with a baseline and week 12 (plus or minus 1 week) assessment that received at least 75% of the planned doses of either etanercept or adalimumab prior to week 12 and who did not have any serious protocol deviations.
Measure: Mean (Standard Deviation); unit: Percentage of B Cells
Arm/Group | Etanercept | Adalimumab
Number analyzed (Participants) | 30 | 18
Percentage of B Cells | 13.2 (7.3) | 13.8 (7.2)
Statistical Analysis 1: Comparison: Etanercept vs Adalimumab; Null Hypothesis: Mean percentage of CD27+ switched memory cells in the peripheral blood at Week 12 does not differ between individuals treated with etanercept and those treated with adalimumab after adjusting for baseline CD27+ switched memory cells. Alt. hypothesis: Mean percentage of CD27+ switched memory cells in the peripheral blood at Week 12 in individuals treated with etanercept is lower than in those treated with adalimumab after adjusting for baseline CD27+ switched memory cells; Test type: Superiority or Other; p = 0.3, ANCOVA; P-value for testing treatment effect uses week 12 CD27+ switched memory as the outcome variable and adjusts for baseline CD27+ switched memory

2. Secondary Outcome: Percentage of Participants Fulfilling DAS-28-CRP "Good or Moderate Response" Criteria at Week 12
Description: Good responders: change in DAS28-CRP (Baseline-Week12) > 1.2 and Week 12 DAS-CRP score was <= 3.2. If the conditions for non-response* or good response were not met, the DAS28-CRP response was considered moderate. Participants with measurements for designated time points were included in the analysis. [*Non-responders had any of 4 conditions: change in DAS28-CRP (Baseline -Week 12) <0.6; 0.6 <= change in DAS28-CRP ( Baseline-Week 12) < 1.2 with Week 12 DAS28-CRP score > 5.1; a flare that required prednisone > 10 mg/day (or equivalent) beyond Week 8 or the inability to taper prednisone to <= 10 mg/day by Week 8; or the participant required prednisone > 20 mg/day at any time point].
Time Frame: Week 12
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either etanercept or adalimumab. Data were not available for two participants who received Etanercept.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Adalimumab
Number analyzed (Participants) | 37 | 19
percentage of participants | 86.5 | 89.5

3. Secondary Outcome: Percentage of Participants Fulfilling DAS-28-CRP "Good or Moderate Response" Criteria at Week 24
Description: Good responders had: change in DAS28-CRP (Baseline-Week 24) > 1.2 and the Week 24 DAS-CRP score was <= 3.2. If the conditions for non-response* or good response were not met then the DAS28-CRP response was considered moderate.[*Non-responders had any of the 4 conditions: change in DAS28-CRP (Baseline -Week 24) <0.6; 0.6 <= change in DAS28-CRP ( Baseline-Week 24) < 1.2 with Week 24 DAS28-CRP score > 5.1 ; a flare that required prednisone > 10 mg/day (or equivalent) beyond Week 8 or the inability to taper prednisone to <= 10 mg/day by Week 8; or the participant required prednisone > 20 mg/day at any time point]. Participants with measurements for designated time points were included in the analysis.
Time Frame: Week 24
Population: The Modified Intent-to-Treat with available data population included all randomized subjects who received at least one dose of either etanercept or adalimumab. Data were not available for five participants who received Etanercept.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Adalimumab
Number analyzed (Participants) | 34 | 19
percentage of participants | 88.2 | 84.2

4. Secondary Outcome: Percentage of Participants Meeting ACR20 Response Criteria at Week 12
Description: The American College of Rheumatology (ACR) 20 Responder Index is defined as someone who achieved at least 20% improvement in the tender and swollen 28-joint count, and 20% improvement in at least three of the following 5 measures:
  * Patient's pain assessment (Visual Analogue Scale (VAS) 100 mm)
  * Patient's global assessment of disease activity (VAS 100 mm)
  * Physician's global assessment of disease activity (VAS 100 mm)
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score)
  * Acute phase reactant (CRP).
  Participants with measurements for designated time points were included in the analysis.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Adalimumab
Number analyzed (Participants) | 37 | 19
percentage of participants | 67.6 | 73.7

5. Secondary Outcome: Percentage of Participants Meeting ACR20 Response Criteria at Week 24
Description: as for outcome 4
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Adalimumab
Number analyzed (Participants) | 34 | 19
percentage of participants | 73.5 | 84.2

6. Secondary Outcome: Percentage of Participants Meeting ACR50 Response Criteria at Week 12
Description: The American College of Rheumatology (ACR) 50 Responder Index is defined as someone who achieved at least 50% improvement in the tender and swollen 28-joint count, and 50% improvement in at least three of the following 5 measures:
  * Patient's pain assessment (Visual Analogue Scale (VAS) 100 mm)
  * Patient's global assessment of disease activity (VAS 100 mm)
  * Physician's global assessment of disease activity (VAS 100 mm)
  * Patient self-assessed disability (Health Assessment Questionnaire (HAQ) score)
  * Acute phase reactant (CRP).
  Participants with measurements for designated time points were included in the analysis.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Adalimumab
Number analyzed (Participants) | 37 | 19
percentage of participants | 29.7 | 47.4

7. Secondary Outcome: Percentage of Participants Meeting ACR50 Response Criteria at Week 24
Description: as for outcome 6
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Adalimumab
Number analyzed (Participants) | 34 | 19
percentage of participants | 38.2 | 63.2

ADVERSE EVENTS:
Time Frame: From the time of administration of the first dose of study drug until the participant completed study participation, an average of 24 weeks, or until 30 days after the participant prematurely withdrew.
Arm/Group | Etanercept | Adalimumab
Serious Adverse Events (participants affected / at risk) | 2/39 | 1/19
Other Adverse Events (participants affected / at risk) | 31/39 | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=39) | Adalimumab (N=19)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=39) | Adalimumab (N=19)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 4 (7) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5) | 3 (5)
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 4 (4) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (9) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 10 (12) | 3 (3)
Blood creatinine increased (Investigations) | 5 (6) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No